CLINICAL TRIAL: NCT04128098
Title: Frequency of Correct Response and Factors Associated in the Medium Term With a Multimodal Rehabilitation Program for Chronic Low Back Pain
Acronym: FRELOMB
Status: Terminated | Type: Observational
Why Stopped: The Covid pandemic made it impossible to monitor and rehabilitate patients at the Dijon Bourgogne CHU's CCR. A new home rehabilitation programme was set up.
  This new rehabilitation programme rendered the study obsolete and the project was abandoned.
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: ORNETTI PCA 2018-2
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation — * Functional tests: 400-meter walking test, 200-meter brisk walking test, Sorensen test, Shirado test, measurement of maximum isometric force of extensors/back flexors.
  * 3D analysis of locomotion and posture
  * Test of the flexion-relaxation phenomenon of the lumbar erector muscles
Other: Questionnaires — Self-questionnaires: Oswestry, Québec, SF-12, VAS pain, HAD, pain dramatization questionnaire, physical activity questionnaires, VAS and GPE satisfaction, FABQ, GPE functional status and EPICES score.
Other: Rehabilitation care program — * Personalized global exercises (aerobics) on ergometers
  * Muscle strengthening with resistance
  * Balneotherapy
  * Learning health skills related to their condition (therapeutic education)
  * Personal and group motivational interviews
  * Nutritional advice
  * Relaxation session

SUMMARY:
Non-specific chronic low back pain is defined as pain that originates in the lumbar spine, is persistent, lasts more than 3 months, and is unrelated to an inflammatory, traumatic, tumour, malformation, or infectious cause. Chronic low back pain is one of the most frequent reasons for consulting a physician, and one of the most common sources of disability, particularly as a result of socio-professional withdrawl. It is a major consumer of health resources (diagnostic investigations, multiple treatments) and involves heavy expenses for the investigator's health insurance system. In view of this major public health issue, in November 2017, the Health Insurance and several specialized health organizations launched a "general public" campaign to raise awareness of low back pain. This campaign, entitled "Back pain? The right treatment is movement" was designed to encourage appropriate physical activity in patients with low back pain.

Among the available therapies, multimodal programs are recommended as a first line treatment. In order to incorporate physical activity into patients' daily lives, these rehabilitation programs are based on a comprehensive multidisciplinary approach (therapeutic education, muscle strengthening, reconditioning, ergonomics, psychological, social, professional and nutritional management and cardiovascular risk factors). Although such programmes have already shown short term effectiveness, few data are available on their continued effectiveness in the medium term (1 year). This project aims to identify good and bad responders to a multimodal program in the medium term, based on common clinical parameters (Quebec City questionnaire score and spontaneous walking speed), and to identify the mechanisms underlying this response.

In addition, in clinical practice, heterogeneity in maintaining the effectiveness of the program is observed but little documented. The limited data available show a heterogeneity of these programs and one of the objectives of this project will be to identify the existing barriers and levers available to improve this situation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Having provided oral consent
* Chronic non-specific low back pain (HAS2015 criteria)
* Eligible for a rehabilitation program
* Patient affiliated or benefiting from a social security scheme

Exclusion Criteria:

* Adult unable to provide consent
* Lumbar spine surgery scheduled in the coming year
* Associated pathologies other than spinal (orthopedic, neurological, vascular, cardiac...) that can affect locomotion
* Root damage with motor deficit <3
* Altered comprehension skills making self-assessment impossible
* Patient subject to a protective measure (guardianship, curatorship)
* Patient subject to a judicial protection
* Pregnant, parturient or breastfeeding woman
* Not fluent in French
* Patient who has already completed a multimodal rehabilitation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient presenting for consultation in the re-education and rehabilitation department of the CHU Dijon Bourgogne
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Proportion of good medium-term responders in a multimodal rehabilitation program | M13 (12 months after the end of the program)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France